CLINICAL TRIAL: NCT00655109
Title: A Comparison of Olopatadine Versus Fluticasone Nasal Spray in the Prevention of the Signs and Symptoms of Allergic Conjunctivitis
Brief Title: A Comparison of Olopatadine and Fluticasone in Patients With Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Greiner, Jack V., OD DO PhD (Individual)
Responsible Party: Jack V. Greiner, OD DO PhD, Ophthalmic Research Associates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-003-04
Record Dates: First submitted 2008-04-02; First posted 2008-04-09 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Conjunctivitis, Allergic
Keywords: Allergic conjunctivitis; Allergic rhinoconjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride; Fluticasone; Sodium Chloride; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Olopatadine
  Interventions: Drug: Olopatadine
- 2 (Active Comparator): Fluticasone
  Interventions: Drug: Fluticasone
- 3 (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Saline
- 4 (Placebo Comparator): Placebo Eyedrops
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Olopatadine — Ophthalmic solution
  Arms: 1
Drug: Fluticasone — Nasal spray
  Arms: 2
Drug: Saline — Nasal spray
  Arms: 3
Drug: Artificial tears — Ophthalmic Solution
  Arms: 4

SUMMARY:
To compare the clinical efficacy of olopatadine and fluticasone in a 3-week single center, double-masked, randomized, placebo controlled parallel treatment conjunctival allergen challenge (CAC) study in patients with allergic conjunctivitis

DETAILED DESCRIPTION:
Study will evaluate the efficacy of nasal anti-allergic therapy compared to ocular anti-allergic therapy in the prevention of ocular allergic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age & either sex, any race
* Willing and able to follow all instructions and attend all study visits
* Positive history of ocular allergies
* Reproducible positive ocular allergic reaction induced by conjunctival allergen challenge

Exclusion Criteria:

* Have planned surgery during trial period
* Female currently pregnant, planning a pregnancy, or lactating
* Use of disallowed medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Ocular itching | Minutes following CAC

SECONDARY OUTCOMES:
Ocular redness | Minutes following CAC

CONTACTS AND LOCATIONS:
Overall Officials: Jack V Greiner, OD, DO, PhD, Principal Investigator — ORA, Inc.
Locations (1):
- Ophthalmic Research Associates, Inc, North Andover, Massachusetts, United States